CLINICAL TRIAL: NCT02821507
Title: A Phase 2, Single Arm, Multi Center Trial Evaluating the Efficacy of the COmbination of Sirolimus and cYclophosphamide in Metastatic or Unresectable Myxoid Liposarcoma and chOndrosarcoma
Brief Title: Sirolimus and Cyclophosphamide in Metastatic or Unresectable Myxoid Liposarcoma and Chondrosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, HansGelderblom, Prof A.J. Gelderblom, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COSYMO
Record Dates: First submitted 2016-01-09; First posted 2016-07-01 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Conventional Chondrosarcoma; Myxoid Liposarcoma; Mesenchymal Chondrosarcoma; Dedifferentiated Chondrosarcoma
MeSH Terms: conditions — Liposarcoma, Myxoid; Chondrosarcoma, Mesenchymal | interventions — Sirolimus; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sirolimus and cyclophosphamide (Experimental): combining sirolimus 4mg daily orally and cyclophosphamide 200mg day 1 to 7 and 15 to 21 orally in a 4 week schedule
  Interventions: Drug: sirolimus and cyclophosphamide

INTERVENTIONS:
Drug: sirolimus and cyclophosphamide

SUMMARY:
Chondrosarcoma and liposarcoma consists of different subtypes with a wide range of patient survival. Current treatment options consist of wide surgical resection, however for patients with a local recurrence or metastatic disease the outcome is poor. New treatment options being evaluated and mouse models show in vivo that mammilian target of rapamycin (mTOR) inhibition can prevent tumour growth. mTOR is an kinase that is present in two complexes and thereby activates multiple pathways. Aberrant mTOR signalling is known to be involved in cancer cell survival. Several clinical studies for patients with bone or soft tissue sarcoma treated with mTOR inhibitors have been conducted and they show promising results. From these studies the investigators can conclude that the combination of an mTOR inhibitor with cyclophosphamide shows promising results in chondrosarcoma. With the lack of other treatment options for unresectable and metastatic chondrosarcoma or myxoid liposarcoma the Eurosarc consortium (www.eurosarc.eu) decided to treat these patients in a standardised way according to a common protocol with the combination of sirolimus and cyclophosphamide using the growth modulation index for evaluation in the current clinical study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven conventional chondrosarcoma
* Or pathologically proven myxoid liposarcoma with PIK3CA mutation or Phosphatase and tensin homolog (PTEN) loss
* Or pathologically proven mesenchymal or dedifferentiated chondrosarcoma
* Patient is 18 years and up
* Documented radiographic progression of disease according to RECIST 1.1 criteria in last 6 months
* Written signed informed consent
* Adequate bone marrow function (Hb ≥ 6.0 mmol/L, absolute neutrophil count ≥ 1.5 x 109/L, platelets ≥ 80 x 109/L)
* Availability of archival tumor material for central review or be able to perform a 3 core fresh biopsy
* Ability to adhere to the study visits and all protocol requirements

Exclusion Criteria:

* Previously treated with an mTOR inhibitor
* Known to be allergic to cyclophosphamide
* Life expectancy of less than 3 months
* No measurable lesions according to RECIST 1.1
* Eastern cooperative oncology group (ECOG) Performance status >2
* Major surgery less than 4 weeks prior to start of treatment
* Known human immunodeficiency virus (HIV) positivity
* A decreased renal function with calculated glomerular filtration rate (GFR) < 30ml/min
* Systemic anti-cancer therapy within 28 days prior to the first dose of study drug , or radiotherapy to a target lesion within 21 days prior to the first dose of study drug
* Pregnant or lactating women
* Other invasive malignancies diagnosed within the last 5 years, except non-melanoma skin cancer and localised cured prostate and cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
The time to progression after start of treatment combination treatment of sirolimus and cyclophosphamide | 16 weeks

SECONDARY OUTCOMES:
Comparing pre-treatment tumor material and tumor material taken during treatment using immunohistochemistry to compare activation of the pS6, Bcl-2 and mTor pathway and DNA analysis for taqman analysis to search for hotspot mutations. | 8 weeks
Register adverse events to evaluate the patient safety and tolerability of the sirolimus and cyclophosphamide combination in myxoid liposarcoma and chondrosarcoma | every 8 weeks until progression (average of 1 year)
To evaluate the response according to response evaluation criteria in solid tumors (RECIST) 1.1 | every 8 weeks until progression (average of 1 year)
Using the growth modulation index (GMI) to evaluate treatment efficiency | every 8 weeks until progression (average of 1 year)
  GMI: Time to progression during sirolimus/cyclophosphamide treatment (TTP2) divided by time to progression before start of this treatment TTP1
The overall survival after start of treatment till death | every 8 weeks until progression (average of 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gelderblom, Prof, Principal Investigator — Leiden University Medical Center
Locations (7):
- LUMC, Leiden, Netherlands
- Spain (6):
  - Hospital de Sant Pau, Barcelona
  - Hospital Val d'Hebron, Barcelona
  - CIO Clara Campal, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario y Politécnico de La Fe, Valencia
  - Instituto Valenciano de Oncología, Valencia